CLINICAL TRIAL: NCT02329444
Title: Remote Ischemic Preconditioning for the Prevention of Contrast-induced Acute Kidney Injury in Diabetic Patients Undergoing Percutaneous Coronary Intervention
Brief Title: The Effect of Remote Ischemic Preconditioning on Elective Percutaneous Coronary Intervention in Diabetic Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Prof Eun-Seok Shin, MD. PhD., Interventional Cardiologist MD. PhD., Ulsan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-08-074
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Contrast Induced Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote Ischemic Preconditioning (Experimental): Patients treated with Remote Ischemic Preconditioning
  Interventions: Procedure: Remote ischemic preconditioning
- Sham ischemic preconditioning (Active Comparator): Patients treated with sham ischemic preconditioning
  Interventions: Procedure: Sham ischemic preconditioning

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — Appropriately sized sphygmomanometer cuff placed around right upper arm; where contraindicated, left arm, with inflation of the cuff up to 200mmHg for 5 minutes, followed by deflation of 5 minutes to allow reperfusion with cycle repeated 3 times.
  Arms: Remote Ischemic Preconditioning
Procedure: Sham ischemic preconditioning — Appropriately sized sphygmomanometer cuff placed around right upper arm; where contraindicated, left arm, with inflation of the cuff up to 50mmHg for 5 minutes, followed by deflation of 5 minutes to allow reperfusion with cycle repeated 3 times.
  Arms: Sham ischemic preconditioning

SUMMARY:
Contrast-induced acute kidney injury (CI-AKI) is a significant iatrogenic complication of contrast media use associated with prolonged hospitalization, cardiovascular events, persistent kidney damage and increased risk of all-cause mortality. When remote ischemic preconditioning is applied before percutaneous coronary intervention (PCI), the kidneys can be protected against ischemia-reperfusion injury and subsequently CI-AKI. In this randomised controlled trial, diabetic nephropathy patients undergoing PCI as part of their assessment and treatment of cardiovascular disease are randomized to receive RIPC or control sham preconditioning.

DETAILED DESCRIPTION:
Contrast-induced acute kidney injury (CI-AKI) is a significant iatrogenic complication of contrast media use associated with prolonged hospitalization, cardiovascular events, persistent kidney damage and increased risk of all-cause mortality. Diabetes with pre-existing renal disease can increase the risk of CI-AKI. Remote ischemic preconditioning (RIPC) is a non-pharmacological strategy inducing transient episodes of ischemia by the occlusion of blood flow in non-target tissue such as a limb, before a subsequent prolonged ischemia-reperfusion injury occurs in a more distant organ. These brief, repeated ischemic episodes in the limb can confer a protection at more remote sites such as the heart, brain, lung, kidney, intestine or skeletal muscle. In a recent pilot study, using RIPC prior to coronary angiography in high risk patients with moderate chronic kidney disease, the authors found that RIPC significantly reduced the incidence of CI-AKI (Er et al Circulation. 2012;126(3),296). We hypothesized that RIPC would be protective as an adjunctive therapy in reducing the incidence of CI-AKI in diabetics with pre-existing CKD. This prospective study was performed to evaluate the efficacy of RIPC for the prevention of CI-AKI among diabetic nephropathy patients undergoing percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent
* All of the following:
* Known diagnosis of Type 2 diabetes
* NSTEMI, unstable or stable angina
* Patients undergoing elective coronary angiography and/or percutaneous coronary intervention
* eGFR < 60 mls/min or ACR > 300 mg/dl

Exclusion Criteria:

* STEMI
* decompensated heart failure in the preceding 6 months
* patients with underlying end stage renal disease on maintenance dialysis
* recent (in the last 3 months) cerebrovascular disease
* chronic liver disease
* chronic obstructive pulmonary disease
* gastrointestinal bleeding
* acute or chronic infection or malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence of CI-AKI | 48 hours
  defined as a creatinine rise of ≥ 25% or an increase of > 0.5mg/dl from baseline within 48 hours after contrast exposure

SECONDARY OUTCOMES:
Relative change in NGAL levels from baseline | 24 hours
  Defined as a change in serum NGAL value from baseline
Absolute change in NGAL levels from baseline | 24 hours
  Defined as a change in serum NGAL value from baseline
Relative change in serum creatinine from baseline | 72 hours
  Defined as a change in serum value from baseline

OTHER OUTCOMES:
Periprocedural myocardial infarction | 24 hours
  Defined as Trop T or CKMB levels >3 times the upper limit of normal

CONTACTS AND LOCATIONS:
Overall Officials: Eun-Seok Shin, MD., PhD., Principal Investigator — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea

REFERENCES:
- [Derived] Balbir Singh G, Ann SH, Park J, Chung HC, Lee JS, Kim ES, Choi JI, Lee J, Kim SJ, Shin ES. Remote Ischemic Preconditioning for the Prevention of Contrast-Induced Acute Kidney Injury in Diabetics Receiving Elective Percutaneous Coronary Intervention. PLoS One. 2016 Oct 10;11(10):e0164256. doi: 10.1371/journal.pone.0164256. eCollection 2016. PMID 27723839